CLINICAL TRIAL: NCT07109778
Title: Impact of Copper to Zinc Ratio on Outcome of End Stage Renal Disease Patients
Brief Title: Copper to Zinc Ratio in End Stage Renal Disease Patients Outcome
Status: Not yet recruiting | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Kerolles Adel Estawrow Saleh, Resident physician, Minia University
Other Study IDs: Copper to Zinc ratio in ESRD
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: ESRD (End Stage Renal Disease); Control Condition
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESRD patients: 100 patients on maintainance hemodialysis
- Control groub: 50 Healthy individuals

SUMMARY:
The goal of this observational clinical trial is to Study the impact of copper to zinc ratio on the outcome of ESRD patients

DETAILED DESCRIPTION:
End-stage renal disease (ESRD) carries high morbidity and mortality due to cardiovascular complications, highlighting the need for ongoing research. Trace elements as copper (Cu), and zinc (Zn), are essential for physiological functions, enzyme activity, metabolism, and immune defense. In ESRD patients, Cu and Zn imbalances, with a higher Cu/Zn ratio are linked to greater cardiovascular problems. The relationship between the Cu/Zn ratio and clinical outcomes in ESRD needs more exploration

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients including those on maintenance HD

Exclusion Criteria:

* Acute kidney injury or rapidly progressive glomerulonephritis, acute infections or active inflammatory conditions as sepsis and autoimmune diseases, liver cirrhosis (Child-Pugh Class B or C), gastrointestinal disorders as inflammatory bowel disease, malabsorption, history of organ transplantation excluding kidney transplantation who may be included in a separate analysis if sufficient numbers are recruited, receiving total parenteral nutrition, Cu or Zn metabolism disorders as Wilson's disease, vitamin complex supplementation or antioxidants within the past 6 months, recent hospitalization within the past 3 months, recent surgery within 3 months, recent blood transfusion < 3 months, Pregnancy or lactation, Malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: this prospective observational Case control study will enroll a well-characterized cohort of 100 adult patients with ESRD(eGFR <15 mL/min/1.73 m²) , including those undergoing maintenance hemodialysis recruited from nephrology clinics and dialysis unit at Minia University Hospital . The recruited patients will be stratified into two groups;
  1. Dialysis ESRD Group: It will include 100 adult patients with ESRD stage 5D on maintenance hemodialysis for at least 6 months.
  2. control groub study the impact of Cu/Zn ratio on outcomme of ESRD patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
To determine whether an elevated serum Cu/Zn ratio is associated with an increased risk of cardiac complications in chronic hemodialysis patients. | 6-8 months
  measuring serum Cu/Zn ratio and determining if it is associated with an increased risk of cardiac complications in chronic hemodialysis patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology and urology hospital, Minia unersity hospital, Faculty of medicine, Minia university, Minya, Egypt

REFERENCES:
- [Background] Xie Y, Liu F, Zhang X, Jin Y, Li Q, Shen H, Fu H, Mao J. Benefits and risks of essential trace elements in chronic kidney disease: a narrative review. Ann Transl Med. 2022 Dec;10(24):1400. doi: 10.21037/atm-22-5969. PMID 36660676
- [Background] Ruiz-Cabello P, Soriano-Maldonado A, Delgado-Fernandez M, Alvarez-Gallardo IC, Segura-Jimenez V, Estevez-Lopez F, Camiletti-Moiron D, Aparicio VA. Association of Dietary Habits with Psychosocial Outcomes in Women with Fibromyalgia: The al-Andalus Project. J Acad Nutr Diet. 2017 Mar;117(3):422-432.e1. doi: 10.1016/j.jand.2016.09.023. Epub 2016 Nov 24. PMID 27890478
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839
- [Background] Henry JD, Crawford JR. The short-form version of the Depression Anxiety Stress Scales (DASS-21): construct validity and normative data in a large non-clinical sample. Br J Clin Psychol. 2005 Jun;44(Pt 2):227-39. doi: 10.1348/014466505X29657. PMID 16004657
- [Background] Duerksen DR, Laporte M, Jeejeebhoy K. Evaluation of Nutrition Status Using the Subjective Global Assessment: Malnutrition, Cachexia, and Sarcopenia. Nutr Clin Pract. 2021 Oct;36(5):942-956. doi: 10.1002/ncp.10613. Epub 2020 Dec 29. PMID 33373482
- [Background] Devlin N, Pickard S, Busschbach J. The Development of the EQ-5D-5L and its Value Sets. 2022 Mar 24. In: Devlin N, Roudijk B, Ludwig K, editors. Value Sets for EQ-5D-5L: A Compendium, Comparative Review & User Guide [Internet]. Cham (CH): Springer; 2022. Chapter 1. Available from http://www.ncbi.nlm.nih.gov/books/NBK589306/ PMID 36810043
- [Background] Cannas D, Loi E, Serra M, Firinu D, Valera P, Zavattari P. Relevance of Essential Trace Elements in Nutrition and Drinking Water for Human Health and Autoimmune Disease Risk. Nutrients. 2020 Jul 13;12(7):2074. doi: 10.3390/nu12072074. PMID 32668647